CLINICAL TRIAL: NCT05735145
Title: A Prospective Randomized Controlled Trial for Concurrent Chemoradiotherapy Combined With Adjuvant Chemotherapy in the Treatment of Advanced Cervical Cancer at 2018 FIGO Staging
Brief Title: Concurrent Chemoradiotherapy Combined With Adjuvant Chemotherapy Treated Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fourth Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 124502004985979665
Record Dates: First submitted 2022-06-24; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Uterine Cervical Neoplasms; Chemoradiotherapy; Adjuvant Chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Platinum; Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concurrent chemoradiotherapy combined with adjuvant chemotherapy (Experimental): Adjuvant chemotherapy in patients with locally advanced cervical cancer who achieved CR after concurrent chemoradiotherapy
  Interventions: Drug: paclitaxel combined with platinum
- concurrent chemoradiotherapy (Other): Observation of patients with locally advanced cervical cancer who achieved CR after concurrent chemoradiotherapy
  Interventions: Drug: paclitaxel combined with platinum

INTERVENTIONS:
Drug: paclitaxel combined with platinum — Adjuvant chemotherapy with paclitaxel combined with platinum
  Other Names: Adjuvant chemotherapy with paclitaxel combined with platinum

SUMMARY:
This study carried out a prospective, randomized, controlled clinical study under the background of intensity-modulated radiation therapy and three-dimensional afterloading therapy. By comparing simultaneous intensity-modulated radiotherapy and chemotherapy combined with adjuvant chemotherapy and simultaneous intensity-modulated radiotherapy and chemotherapy alone, based on the 2018 FIGO staging The clinical efficacy of locally advanced cervical cancer further clarifies the role of adjuvant chemotherapy in locally advanced cervical cancer.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the standard treatment for locally advanced cervical cancer, but there are still many patients with local recurrence or metastasis after treatment, and the 5-year survival rate is low. Concurrent chemoradiotherapy followed by adjuvant chemotherapy for locally advanced cervical cancer is still controversial in improving disease-free survival and overall survival, and previous studies were mostly based on traditional two-dimensional radiotherapy techniques, intensity-modulated radiotherapy and three-dimensional afterloading in dosimetry and radiotherapy. Compared with traditional radiotherapy, it has more advantages in terms of biological effects. In addition, after the adjustment of the new 2018 FIGO staging, it is possible to change the impact of the original treatment mode on overall survival. Therefore, more evidence-based medical evidence is needed to clarify the clinical value of adjuvant chemotherapy in the treatment of locally advanced cervical cancer. Therefore, this study carried out a prospective, randomized, controlled clinical study under the background of intensity-modulated radiation therapy and three-dimensional afterloading therapy. By comparing simultaneous intensity-modulated radiotherapy and chemotherapy combined with adjuvant chemotherapy and simultaneous intensity-modulated radiotherapy and chemotherapy alone, based on the 2018 FIGO staging The clinical efficacy of locally advanced cervical cancer further clarifies the role of adjuvant chemotherapy in locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer confirmed by histopathology incloud squamous cell carcinoma, adenocarcinoma and adenosquamous carcinoma
* FIGO stage IB3, IIA2, IIB-IVA patients in 2018
* Locally advanced cervical cancer patients received standard concurrent intensity-modulated chemoradiotherapy followed by three-dimensional afterloading treatment after diagnosis, and the effect reached CR after treatment
* Aged 18-75 years
* PS score 0-1
* Serum hemoglobin >=100*10^9/L, blood platelet >= 100000/μL, absolute count of neutrophils>=1500/μL; 7.Serum creatinine <=1.5 UNL or creatinine clearance >= 60 ml/min; 8.Serum bilirubin <=1.5 UNL, AST (SGOT) and ALT (SGPT)<= 1.5 UNL
* Sign a formal informed consent to show that they understand that the study is in line with hospital and national policies .Estimated total survival > 6 months.

Exclusion Criteria:

* Locally advanced cervical cancer patients received standard concurrent intensity-modulated chemoradiotherapy followed by three-dimensional afterloading treatment after diagnosis, and the effect unreached CR after treatment
* Patients who have received neoadjuvant chemotherapy and surgery
* Patients with cognitive impairment
* Patients with any distant metastases
* Patients with any other malignancy within 5 years
* Any other disease or condition is contraindications to chemoradiotherapy (e.g., active infection, 6 months after myocardial infarction, symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmias, immunosuppressive therapy, etc.); 5.Pregnant or lactating women, or fertile women who do not use contraception
* Severe bone marrow dysfunction
* Patients with bleeding tendency
* Drug abusers or alcohol addicts
* Those who are known to have a third or fourth degree allergic reaction to any treatment in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — femal
Enrollment: 108 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Refers to the time from randomization to the first occurrence of disease progression or death from any cause，whichever came first, assessed up to 1000 months
  progression-free survival

SECONDARY OUTCOMES:
OS | Refers to the time from randomization to death from any cause, assessed up to 1000 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Feng chengjun, Principal Investigator — The The Fourth Affiliated Hospital of Guangxi Medical University
Locations (1):
- the Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi, China